CLINICAL TRIAL: NCT06648603
Title: Citizen Action for Sustainable Dengue Control in Sub-Saharan Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Centre Suisse de Recherches Scientifiques en Cote d'Ivoire (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: C21047
Record Dates: First submitted 2024-07-01; First posted 2024-10-18 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2023-12

CONDITIONS: Dengue
Keywords: Aedes Aegypti; Vector control; Community based intervention; Participatory research; Dengue; Africa; Ivory Coast
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial with 2x2 factorial design - 40 clusters, 10 clusters per study arm (4 arms)
Who Masked: Outcomes Assessor
Masking Description: Statistician unaware of the arms allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Non-intervened control arm: no community-based larval source management (LSM) or BG-GAT intervention
- Community-based larval source management (Experimental): LSM intervention arm: Aedes larval source reduction carried out by trained and supervised local community members
  Interventions: Behavioral: Community-based larval source management
- Enhanced Aedes adults trapping (BG-GAT) (Experimental): BG-GAT intervention arm: Aedes adult mass trapping by BG-GAT set up and maintained by trained and supervised local community members
  Interventions: Device: Enhanced Aedes adults trapping (BG-GAT)
- Community-based larval source management + Enhanced Aedes adults trapping (BG-GAT) (Experimental): Combined LSM and BG-GAT intervention arm: simultaneous Aedes larval source reduction and Aedes adult mass trapping by BG-GAT carried out by trained and supervised local community members
  Interventions: Combination Product: Community-based larval source management with Enhanced Aedes adults trapping (BG-GAT)

INTERVENTIONS:
Behavioral: Community-based larval source management — This project will foster active engagement with community stakeholders, including healthcare workers, community leaders, and other key informants, through participatory meetings aimed at co-creating and developing larval source reduction measures tailored to community's needs. This method emphasizes a participatory framework, ensuring that interventions are both community-informed and culturally relevant.
  Arms: Community-based larval source management
Device: Enhanced Aedes adults trapping (BG-GAT) — Furthermore, the project intends to determine whether the addition of cost-effective, gravid female mosquito-targeting traps, specifically two Biogents Gravid Aedes Traps (BG-GAT) per household, can improve the overall success of these community-based intervention.
  Arms: Enhanced Aedes adults trapping (BG-GAT)
Combination Product: Community-based larval source management with Enhanced Aedes adults trapping (BG-GAT) — The community-based interventions and the BG-GAT deployment will be evaluated in combination to assess their individual and synergistic effects on vector control. This dual strategy combines local participation and practical, evidence-based solutions to address mosquito-borne illness transmission.
  Arms: Community-based larval source management + Enhanced Aedes adults trapping (BG-GAT)

SUMMARY:
This project focuses on addressing arboviral outbreaks in Ivory Coast by involving local communities in the sustainable control of Aedes mosquitoes, utilizing scientific advice and environmental interventions. It will evaluate the impact of a participatory strategy on decreasing mosquito populations and the risk of virus transmission, aiming to provide insights for policy development on disease prevention.

DETAILED DESCRIPTION:
This project targets the growing threat of Aedes mosquito-borne diseases such as dengue in Africa, focusing on the Anono and Gbagba communities in Abidjan, Ivory Coast, by transitioning from traditional control approaches to a community-driven strategy. It focuses on educating and involving communities in the design of sustainable mosquito management measures, such as breeding site eradication and adult mosquito capturing, with scientific experts guiding the efforts. The approach will entail conducting sociocultural surveys and interactive workshops while also encouraging local participation and multi-sectoral collaboration. A randomized controlled trial (RCT) will test this effectiveness of this novel integrated community-based participatory intervention approach in reducing the transmission of Aedes mosquito and other arboviruses. This effort seeks to develop a scalable model for arboviral disease control, promote community resilience, and inform policy recommendations for better public health outcomes in resource-constrained urban settings.

ELIGIBILITY:
Inclusion criteria:

1. Geographical location: households must be located within the designated clusters in the two districts involved in the trial.
2. Participation in cluster arms: households must belong to a cluster that is assigned to one of the four arms (1. Control, 2. Community-based larval source management, 3 Enhanced Aedes adults trapping (BG-GAT), 4. Enhanced Aedes adults trapping (BG-GAT) + Community-based larval source management).
3. Willingness to participate: households agreed to allow researchers to place mosquito traps and conduct larval and adult mosquito surveys.
4. Socio-Environmental Data: households must agree and provide consent to participate to the socio-environmental questionnaire.

Exclusion Criteria:

1. Outside of trial clusters: households located outside the designated clusters in the two districts were excluded.
2. Refusal to participate: households that do not consent to mosquito trap placement or surveys
3. Inaccessibility: households that are not accessible for regular visits or data collection (e.g., due to relocation or difficult terrain).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Aedes aegypti mean number per trap per day | Continuously during months 1-4 (baseline) and months 5-17 (trial)
  Biting rate is the mean number of Aedes females per trap and per day. The proportion of unfed, fed, half-gravid and gravid females will be estimated.

SECONDARY OUTCOMES:
House index | Before (month 1), twice during (month 4, 8) and once at the end of the trial (month 12)
  House index: proportion of houses with at least one larva
Pupal indices: pupae per person index, pupa index and pupae per hectare index | Before (month 1), twice during (month 4, 8) and once at the end of the trial (month 12)
  Pupae per person index: number of pupae per person Pupa index: number of pupae per house Pupae per hectare index: number of pupae per ha
Adults: parity rate | Continuously during months 1-4 (baseline) and months 5-17 (trial)
  The parity rate (PR) (proposition of parous females) will be calculated to estimate vector longevity.
Knowledge, attitudes, and practices on Dengue prevention among the population of Cocody-Bingerville | Before (month 1) the start of the trial and at the end of the trial (month 12)
  A Knowledge, Attitudes, and Practices (KAP) study will be conducted to assess the communities' understanding, attitudes, practices, and beliefs related to dengue. This will be done using a structured questionnaire developed specifically for this trial. The questionnaire comprises both multiple-choice and open-ended questions, allowing for a comprehensive assessment of: 1) Knowledge: Understanding of dengue transmission, symptoms, and prevention, 2) Attitudes: Perceptions of dengue risk and confidence in prevention methods, 3) Practices: Reported behaviors to prevent dengue, such as mosquito control measures. This structured tool will be used at both baseline and endline to measure changes and assess the effectiveness of the intervention."
Mapping and describe Aedes aegypti breeding sites, focusing on their geographic and ecological characteristics. This mapping will be used to enhance targeted larval control efforts in these areas. | Before (month 1) the start of the trial and at the end of the trial (month 12)
  The geographic survey will collect household and environmental data, including demographic details, public space quality, water provision, sanitation access, and waste management practices. It will map housing conditions, examining building types, construction materials, and key features like water storage and solid waste management. The survey will also assess local built environments to inform interventions for improving living conditions and controlling mosquito breeding sites.
Container index | before (month 1), twice during (month 4, 8) and once at the end of the trial (month 12)
  Proportion of positive containers
Breteau index | Before (month 1), twice during (month 4, 8) and once at the end of the trial (month 12)
  Number of positive containers per 100 houses

CONTACTS AND LOCATIONS:
Overall Officials: Pie Müller, PD, PhD, Principal Investigator — Swiss Tropical & Public Health Institute
Locations (1):
- Centre Suisse de Recherches Scientifiques en Côte d'Ivoire, Abidjan, Côte d’Ivoire

IPD SHARING:
Plan to Share IPD: No